CLINICAL TRIAL: NCT01131559
Title: Adjunctive Lisdexamfetamine in Bipolar Depression
Brief Title: Adjunctive Lisdexamfetamine (LDX) in Bipolar Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor halted study.
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Shire (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adjunctive LDX in BP
Record Dates: First submitted 2010-03-19; First posted 2010-05-27 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar; Depression
Keywords: bipolar disorder; manic depression; depression; Bipolar I or II
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine (Active Comparator): Drug
  Interventions: Drug: Lisdexamfetamine
- Placebo (Placebo Comparator): Drug
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Lisdexamfetamine — Oral; 20-70mg/day
  Other Names: Vyvanse
  Arms: Lisdexamfetamine
Drug: Placebo control — Oral; 20-70mg/day
  Other Names: Sugar pill, fake pill with no active medication
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the efficacy and tolerability of lisdexamfetamine in the adjunctive treatment of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet DSM-IV-TR criteria bipolar I or II disorder,

Exclusion Criteria:

* Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease. Subjects should be biochemically euthyroid to enter the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in MADRS score | 30-36 months
  The primary efficacy variable is baseline-to-endpoint change in Montgomery-Asberg Depression Rating Scale (MADRS) score.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- See also: Link to facility where study is conducted — http://lindnercenterofhope.org/research